CLINICAL TRIAL: NCT07021313
Title: Deliver mOre aPplications for More Durable Pulmonary Vein IsOlation
Acronym: DOPPIO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: R&D Cardiologie (Other)
Responsible Party: Principal Investigator, L.V.A. Boersma, Clinical professor, R&D Cardiologie
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL88354.100.24
Record Dates: First submitted 2025-05-30; First posted 2025-06-13 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Atrial Fibrillation
Keywords: Pulsed Field Ablation; Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in a 1:1 fashion with a block size of 4 to the study arm or the usual care (control) arm.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Experimental arm, extra applications (Experimental): Pulmonary vein isolation will be performed with the pentaspline ablation catheter in an olive-shape (2x), basket shape (4x), and flower shape (6x) at each vein
  Interventions: Device: Pulmonary vein isolation by percutaneous endocardial catheter ablation using the FARAPULSE pulsed high voltage electrical field system in patients with atrial fibrillation
- Control arm, standard of care (Active Comparator): Pulmonary vein isolation will be performed with the pentaspline catheter in basket shape (4x) and flower shaped (4x) applications of the catheter.
  Interventions: Device: Pulmonary vein isolation by percutaneous endocardial catheter ablation using a pentaspline pulsed high voltage electrical field system in patients with atrial fibrillation

INTERVENTIONS:
Device: Pulmonary vein isolation by percutaneous endocardial catheter ablation using the FARAPULSE pulsed high voltage electrical field system in patients with atrial fibrillation — Standard of care 4 pulsed electrical field applications in basket shape and 4 applications in flower shape
  Arms: Experimental arm, extra applications
Device: Pulmonary vein isolation by percutaneous endocardial catheter ablation using a pentaspline pulsed high voltage electrical field system in patients with atrial fibrillation — Experimental treatment delivering 2 pulsed electrical field applications in olive shape, 4 in basket shape and 6 applications in flower shape
  Arms: Control arm, standard of care

SUMMARY:
Pulmonary vein isolation (PVI) by catheter ablation (CA) has become a widely accepted interventional treatment for patients with symptomatic atrial fibrillation (AF) despite anti-arrhythmic drugs (AAD). Classic thermal ablation modalities use radiofrequency energy or cryo-energy to create cardiac tissue lesions. Irreversible electroporation (IRE) using pulsed field energy (PFA) is a novel technology for cardiac tissue ablation. Initial studies have shown favorable outcome data in patients with AF treated by performing PVI using PFA. However, the freedom of AF has not yet proven superior to existing thermal ablation methods and appears similarly associated with suboptimal lesion durability, leading to electrical reconnection. The purpose of this study is to determine if freedom of atrial fibrillation may be improved by delivering more and better targeted pulsed field ablations.

DETAILED DESCRIPTION:
Pulmonary vein isolation (PVI) by catheter ablation (CA) has become a widely accepted interventional treatment for patients with symptomatic atrial fibrillation (AF) despite anti-arrhythmic drugs (AAD). Classic thermal ablation modalities use radiofrequency energy or cryo-energy to create cardiac tissue lesions. Irreversible electroporation (IRE) using pulsed field energy (PFA) is a novel technology for cardiac tissue ablation. Initial studies have shown favorable outcome data in patients with AF treated by performing PVI using PFA. However, the freedom of AF has not yet proven superior to existing thermal ablation methods and appears similarly associated with suboptimal lesion durability, leading to electrical reconnection. The purpose of this study is to determine if freedom of atrial fibrillation may be improved by delivering more and better targeted pulsed field ablations. Patients will undergo the standard catheter ablation procedure in accordance with good clinical practice, performing pulmonary vein islolation (PVI) with the FARAPULSE cardiac ablation system. In the control group PVI will be performed with 4 basket- and 4 flower-shaped applications of the catheter, while in the study group 2 olive-, 4 basket-, and 6 flower shaped applications will be delivered at each vein. All other procedural steps will be the same between groups. Patients will be randomized in a 1:1 fashion with a block size of 4 to the study arm or the usual care (control) arm. The primary study parameter for efficacy is the freedom of atrial arrhythmias after the 2-month blanking period up to 12 months after the procedure. The secondary study outcomes include the extent and position of pulmonary vein reconnection observed during redo procedures that are performed due to arrhythmia recurrence, which constitutes a study endpoint. Furthermore, the study also evaluates arrhythmia burden after the procedure in centers that routinely use photoplethysmographic remote monitoring as standard care for all their ablation patients.

ELIGIBILITY:
Inclusion Criteria:

* Be scheduled for PVI with the use of the FARAPULSE catheter ablation system AND
* Have paroxysmal atrial fibrillation (PAF) documented in the last 6 months prior to enrolment OR
* Had persistent atrial fibrillation but maintained in SR or converted to paroxysmal by antiarrhythmic drugs with no more than 1 cardioversion beyond 7 days in the past

Exclusion Criteria:

* Cerebrovascular accident (CVA) in the last 6 months
* More than moderate valvular disease that would require intervention
* Cardiac catheter/surgical intervention in the last 3 months or scheduled
* Atrial septal defect (ASD)/ patent foramen ovale (PFO) closure in the past
* Left atrial appendage (LAA) closure in the past
* Mechanical mitral valve
* Non-adherence to oral anticoagulation in the 3 weeks prior to ablation
* Renal disease with known eGFR<45 ml
* Left atrial volume index (LAVI) >50 ml/m2 or left atrial diameter (LAD) >50 mm
* Known contra-indication for catheter ablation
* Known contra-indication for deep sedation or general anesthesia
* Known pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Freedom of atrial fibrillation after a 2-month blanking period up to 12 months post procedure. | Baseline, month 3, month 6, month 12.
  The primary efficacy outcome will be the freedom of arrhythmias lasting >30 seconds after a single PVI ablation procedure from the blanking period of 2 months until 12 months follow-up after ablation.
  The use of class I or III antiarrhythmic drugs should be stopped at the 3-month visit at the end of the blanking period, or else will count as treatment failure.
  Any left-sided ablation procedure after a successful index procedure will count as treatment failure.
  An atrioventricular (nodal) reentry tachycardia (AVNRT/AVRT), or typical right atrial flutter occurring after the index procedure, will not count as treatment failure.

SECONDARY OUTCOMES:
Procedural-up-to-30 days and 30 days up-to 12 months safety of increasing PFA application numbers | From procedure to 12-month follow-up
  Compare the number of major adverse event between both study arms including (but not exclusively) cardiac tamponade, clinically relevant pulmonary vein stenosis, atrio-esophageal fistula, stroke, persisting phrenic nerve palsy, major bleeding (BARC criteria), hemolysis, cardiac arrest, death
Quality of life differences between groups | Baseline, month 3, month 6, month 12.
  QOL will be assessed with the Atrial Fibrillation Quality of Life Questionaire scoring system asking 18 question with a score on a scale of 1-7 and a range of 0-100. This will be compared between both study arms
The potential for hemolysis in relation to application number | Post procedure every 24 hours, up to 5 days post procedure for each individual patient
  Hemolysis will be assessed by testing urine-samples with hemosticks based on the grading system of the urine stick. In case of a positive urine-stick patients will undergo further diagnostic testing by blood test to determine severity of hemolysis. The number patients with hemolysis and the severity of hemolysis between the study arms will be evaluated
The durability of pulmonary vein isolation in case of a redo procedure | Month 3, month 6, month 12.
  Mapping of the electrical activity of each pulmonary vein will performed in each patient undergoing a repeat ablation procedure. The number and pattern of electrical reconnection will be compared between both study arms

CONTACTS AND LOCATIONS:
Overall Officials: Lucas VA Boersma, MD, PhD, Principal Investigator — St. Antonius Hospital
Locations (1):
- St. Antonius Hospital, Nieuwegein, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Boersma L, Andrade JG, Betts T, Duytschaever M, Purerfellner H, Santoro F, Tzeis S, Verma A. Progress in atrial fibrillation ablation during 25 years of Europace journal. Europace. 2023 Aug 2;25(9):euad244. doi: 10.1093/europace/euad244. PMID 37622592
- [Background] Kawamura I, Neuzil P, Shivamurthy P, Kuroki K, Lam J, Musikantow D, Chu E, Turagam MK, Minami K, Funasako M, Petru J, Choudry S, Miller MA, Langan MN, Whang W, Dukkipati SR, Koruth JS, Reddy VY. How does the level of pulmonary venous isolation compare between pulsed field ablation and thermal energy ablation (radiofrequency, cryo, or laser)? Europace. 2021 Nov 8;23(11):1757-1766. doi: 10.1093/europace/euab150. PMID 34151947
- [Background] Calkins H, Hindricks G, Cappato R, Kim YH, Saad EB, Aguinaga L, Akar JG, Badhwar V, Brugada J, Camm J, Chen PS, Chen SA, Chung MK, Cosedis Nielsen J, Curtis AB, Davies DW, Day JD, d'Avila A, Natasja de Groot NMS, Di Biase L, Duytschaever M, Edgerton JR, Ellenbogen KA, Ellinor PT, Ernst S, Fenelon G, Gerstenfeld EP, Haines DE, Haissaguerre M, Helm RH, Hylek E, Jackman WM, Jalife J, Kalman JM, Kautzner J, Kottkamp H, Kuck KH, Kumagai K, Lee R, Lewalter T, Lindsay BD, Macle L, Mansour M, Marchlinski FE, Michaud GF, Nakagawa H, Natale A, Nattel S, Okumura K, Packer D, Pokushalov E, Reynolds MR, Sanders P, Scanavacca M, Schilling R, Tondo C, Tsao HM, Verma A, Wilber DJ, Yamane T; Document Reviewers:. 2017 HRS/EHRA/ECAS/APHRS/SOLAECE expert consensus statement on catheter and surgical ablation of atrial fibrillation. Europace. 2018 Jan 1;20(1):e1-e160. doi: 10.1093/europace/eux274. No abstract available. PMID 29016840
- [Background] Koruth J, Verma A, Kawamura I, Reinders D, Andrade JG, Deyell MW, Mehta N, Reddy VY. PV Isolation Using a Spherical Array PFA Catheter: Preclinical Assessment and Comparison to Radiofrequency Ablation. JACC Clin Electrophysiol. 2023 May;9(5):652-666. doi: 10.1016/j.jacep.2023.01.022. Epub 2023 Feb 3. PMID 36842871
- [Background] Futing A, Reinsch N, Howel D, Brokkaar L, Rahe G, Neven K. First experience with pulsed field ablation as routine treatment for paroxysmal atrial fibrillation. Europace. 2022 Jul 21;24(7):1084-1092. doi: 10.1093/europace/euac041. PMID 35513354
- [Background] Verma A, Asivatham SJ, Deneke T, Castellvi Q, Neal RE 2nd. Primer on Pulsed Electrical Field Ablation: Understanding the Benefits and Limitations. Circ Arrhythm Electrophysiol. 2021 Sep;14(9):e010086. doi: 10.1161/CIRCEP.121.010086. Epub 2021 Sep 20. PMID 34538095
- [Background] Reddy VY, Neuzil P, Koruth JS, Petru J, Funosako M, Cochet H, Sediva L, Chovanec M, Dukkipati SR, Jais P. Pulsed Field Ablation for Pulmonary Vein Isolation in Atrial Fibrillation. J Am Coll Cardiol. 2019 Jul 23;74(3):315-326. doi: 10.1016/j.jacc.2019.04.021. Epub 2019 May 11. PMID 31085321
- [Background] Hartl S, Reinsch N, Futing A, Neven K. Pearls and Pitfalls of Pulsed Field Ablation. Korean Circ J. 2023 May;53(5):273-293. doi: 10.4070/kcj.2023.0023. PMID 37161743
- [Background] Reddy VY, Dukkipati SR, Neuzil P, Anic A, Petru J, Funasako M, Cochet H, Minami K, Breskovic T, Sikiric I, Sediva L, Chovanec M, Koruth J, Jais P. Pulsed Field Ablation of Paroxysmal Atrial Fibrillation: 1-Year Outcomes of IMPULSE, PEFCAT, and PEFCAT II. JACC Clin Electrophysiol. 2021 May;7(5):614-627. doi: 10.1016/j.jacep.2021.02.014. Epub 2021 Apr 28. PMID 33933412
- [Background] Reddy VY, Gerstenfeld EP, Natale A, Whang W, Cuoco FA, Patel C, Mountantonakis SE, Gibson DN, Harding JD, Ellis CR, Ellenbogen KA, DeLurgio DB, Osorio J, Achyutha AB, Schneider CW, Mugglin AS, Albrecht EM, Stein KM, Lehmann JW, Mansour M; ADVENT Investigators. Pulsed Field or Conventional Thermal Ablation for Paroxysmal Atrial Fibrillation. N Engl J Med. 2023 Nov 2;389(18):1660-1671. doi: 10.1056/NEJMoa2307291. Epub 2023 Aug 27. PMID 37634148
- [Background] Schmidt B, Bordignon S, Neven K, Reichlin T, Blaauw Y, Hansen J, Adelino R, Ouss A, Futing A, Roten L, Mulder BA, Ruwald MH, Mene R, van der Voort P, Reinsch N, Kueffer T, Boveda S, Albrecht EM, Schneider CW, Chun KRJ. EUropean real-world outcomes with Pulsed field ablatiOn in patients with symptomatic atRIAl fibrillation: lessons from the multi-centre EU-PORIA registry. Europace. 2023 Jul 4;25(7):euad185. doi: 10.1093/europace/euad185. PMID 37379528
- [Background] Verma A, Haines DE, Boersma LV, Sood N, Natale A, Marchlinski FE, Calkins H, Sanders P, Packer DL, Kuck KH, Hindricks G, Onal B, Cerkvenik J, Tada H, DeLurgio DB; PULSED AF Investigators. Pulsed Field Ablation for the Treatment of Atrial Fibrillation: PULSED AF Pivotal Trial. Circulation. 2023 May 9;147(19):1422-1432. doi: 10.1161/CIRCULATIONAHA.123.063988. Epub 2023 Mar 6. PMID 36877118
- [Background] Tohoku S, Chun KRJ, Bordignon S, Chen S, Schaack D, Urbanek L, Ebrahimi R, Hirokami J, Bologna F, Schmidt B. Findings from repeat ablation using high-density mapping after pulmonary vein isolation with pulsed field ablation. Europace. 2023 Feb 16;25(2):433-440. doi: 10.1093/europace/euac211. PMID 36427201
- [Background] Nakatani Y, Sridi-Cheniti S, Cheniti G, Ramirez FD, Goujeau C, Andre C, Nakashima T, Eggert C, Schneider C, Viswanathan R, Krisai P, Takagi T, Kamakura T, Vlachos K, Derval N, Duchateau J, Pambrun T, Chauvel R, Reddy VY, Montaudon M, Laurent F, Sacher F, Hocini M, Haissaguerre M, Jais P, Cochet H. Pulsed field ablation prevents chronic atrial fibrotic changes and restrictive mechanics after catheter ablation for atrial fibrillation. Europace. 2021 Nov 8;23(11):1767-1776. doi: 10.1093/europace/euab155. PMID 34240134
- [Background] Cochet H, Nakatani Y, Sridi-Cheniti S, Cheniti G, Ramirez FD, Nakashima T, Eggert C, Schneider C, Viswanathan R, Derval N, Duchateau J, Pambrun T, Chauvel R, Reddy VY, Montaudon M, Laurent F, Sacher F, Hocini M, Haissaguerre M, Jais P. Pulsed field ablation selectively spares the oesophagus during pulmonary vein isolation for atrial fibrillation. Europace. 2021 Sep 8;23(9):1391-1399. doi: 10.1093/europace/euab090. PMID 33961027
- [Background] Musikantow DR, Neuzil P, Petru J, Koruth JS, Kralovec S, Miller MA, Funasako M, Chovanec M, Turagam MK, Whang W, Sediva L, Dukkipati SR, Reddy VY. Pulsed Field Ablation to Treat Atrial Fibrillation: Autonomic Nervous System Effects. JACC Clin Electrophysiol. 2023 Apr;9(4):481-493. doi: 10.1016/j.jacep.2022.10.028. Epub 2022 Nov 30. PMID 36752473
- [Background] Reddy VY, Petru J, Funasako M, Kopriva K, Hala P, Chovanec M, Janotka M, Kralovec S, Neuzil P. Coronary Arterial Spasm During Pulsed Field Ablation to Treat Atrial Fibrillation. Circulation. 2022 Dec 13;146(24):1808-1819. doi: 10.1161/CIRCULATIONAHA.122.061497. Epub 2022 Sep 22. PMID 36134574
- [Background] Bohnen M, Weber R, Minners J, Jadidi A, Eichenlaub M, Neumann FJ, Arentz T, Lehrmann H. Characterization of circumferential antral pulmonary vein isolation areas resulting from pulsed-field catheter ablation. Europace. 2023 Feb 8;25(1):65-73. doi: 10.1093/europace/euac111. PMID 35852306
- [Background] Haissaguerre M, Jais P, Shah DC, Takahashi A, Hocini M, Quiniou G, Garrigue S, Le Mouroux A, Le Metayer P, Clementy J. Spontaneous initiation of atrial fibrillation by ectopic beats originating in the pulmonary veins. N Engl J Med. 1998 Sep 3;339(10):659-66. doi: 10.1056/NEJM199809033391003. PMID 9725923
- [Background] Patel C, Gerstenfeld EP, Gupta SK, Winterfield J, Woods C, Natale A, Schneider CW, Achyutha AB, Holland SK, Richards E, Albrecht EM, Lehmann JW, Mansour M, Reddy VY. Comparison of cerebral safety after atrial fibrillation using pulsed field and thermal ablation: Results of the neurological assessment subgroup in the ADVENT trial. Heart Rhythm. 2024 Nov;21(11):2103-2109. doi: 10.1016/j.hrthm.2024.05.048. Epub 2024 May 31. PMID 38823667
- [Background] Mansour M, Gerstenfeld EP, Patel C, Natale A, Whang W, Cuoco FA, Mountantonakis SE, Gibson DN, Harding JD, Holland SK, Achyutha AB, Schneider CW, Mugglin AS, Albrecht EM, Stein KM, Lehmann JW, Reddy VY. Pulmonary vein narrowing after pulsed field versus thermal ablation. Europace. 2024 Feb 1;26(2):euae038. doi: 10.1093/europace/euae038. PMID 38305503
- [Background] Reddy VY, Anic A, Koruth J, Petru J, Funasako M, Minami K, Breskovic T, Sikiric I, Dukkipati SR, Kawamura I, Neuzil P. Pulsed Field Ablation in Patients With Persistent Atrial Fibrillation. J Am Coll Cardiol. 2020 Sep 1;76(9):1068-1080. doi: 10.1016/j.jacc.2020.07.007. PMID 32854842
- [Background] du Pre BC, van Driel VJ, van Wessel H, Loh P, Doevendans PA, Goldschmeding R, Wittkampf FH, Vink A. Minimal coronary artery damage by myocardial electroporation ablation. Europace. 2013 Jan;15(1):144-9. doi: 10.1093/europace/eus171. Epub 2012 May 31. PMID 22654094
- [Background] Moshkovits Y, Grynberg D, Heller E, Maizels L, Maor E. Differential effect of high-frequency electroporation on myocardium vs. non-myocardial tissues. Europace. 2023 Feb 16;25(2):748-755. doi: 10.1093/europace/euac191. PMID 36305566
- [Background] Popa MA, Venier S, Mene R, Della Rocca DG, Sacher F, Derval N, Hocini M, Dulucq S, Caluori G, Combes S, Albenque JP, Saitta F, Haller B, Chierchia GB, de Asmundis C, Defaye P, Boveda S, Jais P. Characterization and Clinical Significance of Hemolysis After Pulsed Field Ablation for Atrial Fibrillation: Results of a Multicenter Analysis. Circ Arrhythm Electrophysiol. 2024 Oct;17(10):e012732. doi: 10.1161/CIRCEP.124.012732. Epub 2024 Aug 30. PMID 39212069